CLINICAL TRIAL: NCT05333354
Title: Effectiveness of Delirium Simulation Education on the Self-efficacy and Critical Thinking Skill of Nurses in Intensive Care Unit- Randomized Clinical Trial
Brief Title: Effectiveness of Delirium Simulation Education of Nurses in Intensive Care Unit
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Yu-Ling Chang, assistant professor, Chang Gung Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MOST109-2314-B-182-009-MY3
Record Dates: First submitted 2022-02-16; First posted 2022-04-19 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Self Efficacy; Nursing Caries; Intensive Care Unit Delirium; Simulation of Physical Illness
Keywords: intensive care unit,nurses,delirium,simulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental(simulation education group) (Experimental): The experimental group (simulation teaching group), the content of simulation teaching is based on the simulation model, and includes five important elements: Instructor, student, educational practice, simulation situation design and characteristics, and result that design covering the four stages of learning, concrete experience, reflective observation, abstract conceptualization and action experience, and design lesson plans, which include delirium assessment and delirium risk factor detection. Delirium prevention and management (PADIS guidelines). The main objectives of the teaching plan design of the experimental group are: to be able to confirm delirium by assessment of the Delirium Assessment Scale; to confirm the risk factors by the history taking; to propose treatment and measures according to the assessment results. Secondary goals: Be able to perform handovers.
  Interventions: Other: education strategy
- Control(traditional group) (No Intervention): Nurses in the control group did not receive simulated situational teaching, but received classroom teaching 3 times (once every other week) (delirium assessment, risk factor assessment; PADIS treatment), each session of about 2 hours. In order to avoid inconsistent teaching content, the control group and the experimental group are not to be together in classroom.

INTERVENTIONS:
Other: education strategy — The educational course of the experimental group will last for 6 weeks, including classroom teaching and simulated situational teaching. The classroom teaching will be divided into 3 times, a course of about 2 hours at a time; after the class, simulated situational teaching is also arranged for 4 hours at a time/ Caring for many patients with delirium, and performing related research. The simulated scenario lesson plan plans to design 3 major themes (delirium assessment, delirium risk factors, delirium prevention, each major theme will have 2 scenarios, each The simulation teaching exercise starts with pre-briefing, and after the end, debriefing reflection and discussion with the students.
  Arms: Experimental(simulation education group)

SUMMARY:
Delirium is a common symptom in the intensive care unit, which greatly affects the prognosis of critically ill patients and increases medical costs. Although many studies have implemented preventive measures, they have not been able to significantly improve the prevalence of delirium, because many medical measures devises in the intensive care unit are still necessary for patients. Therefore, early detection of patients with delirium symptoms, risk factors, and immediate Delirium management is important. Nurses are the first line of clinically important roles in assessing delirium symptoms. So, design a delirium simulation education for nurses is important.

DETAILED DESCRIPTION:
Through literature review, the investigators found that research on delirium in the intensive care unit simulated education interventions are insufficient, and longitudinal studies to explore how long the effect can be maintained or delirium assessment and delirium management are designed dependent on theory are lacking. Therefore, the purpose of this study was to investigate the effect of delirium simulation education on delirium knowledge, delirium critical thinking, delirium care self-efficacy and satisfaction among nurses in intensive care units, and to explore the influencing factors.

ELIGIBILITY:
Inclusion Criteria:

1. Nurses who have worked in the intensive care unit for more than 3 months,
2. No physical or mental illness or recent major family events,
3. Never received delirium simulation training.

Exclusion Criteria:

1. Those who are not working in the intensive care unit for less than 3 months,
2. Those who have recently suffered from physical and mental illness or a major family event recently,
3. Those who have received delirium simulation training,
4. Those who are currently working as nursing supervisors.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-08-01 (Estimated); Primary Completion 2023-07-31 (Estimated); Study Completion 2023-07-31 (Estimated)

PRIMARY OUTCOMES:
Effectiveness change of delirium care knowledge after simulation teaching | change from baseline in delirium knowledge and 3, 6, 12 months after intervention
  Effectiveness of participants with simulation teaching as assessed by delirium knowledge questioner, change from baseline in knowledge scores on delirium knowledge questioner at 3,6,12 months
Effectiveness change of delirium care self-efficacy after simulation teaching | change from baseline in delirium care self-efficacy and 3, 6, 12 months after intervention
  Effectiveness of participants with simulation teaching as assessed by delirium care self-efficacy questioner, change from baseline in self-efficacy scores on delirium care self-efficacy questioner at 3,6,12 months
Effectiveness change of delirium critical thinking skills after simulation teaching | change from baseline in delirium critical thinking skills and 3, 6, 12 months after intervention
  Effectiveness of participants with simulation teaching as assessed by delirium critical thinking skills questioner, change from baseline in critical thinking skills scores on delirium critical thinking skills questioner at 3,6,12 months

IPD SHARING:
Plan to Share IPD: No